CLINICAL TRIAL: NCT07404670
Title: A Multicenter, Prospective Study to Analyze the Efficacy and Safety of Microwave Ablation for the Treatment of Vascular Malformations
Brief Title: Microwave Ablation for Treatment of Vascular Malformations: Efficacy and Safety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chunshui He, Ph.D , Chief Physician of Vascular Surgery , Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu University of Traditional Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChengduUTCM VM
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Venous Malformations; Arteriovenous Malformations; Microwave Ablation; Vascular Malformations
Keywords: Microwave Ablation; Vascular Malformations; Venous Malformations; Arteriovenous Malformations; Minimally Invasive Treatment
MeSH Terms: conditions — Arteriovenous Malformations; Vascular Malformations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microwave Ablation for Vascular Malformations (Experimental): Patients in this arm will receive microwave ablation for the treatment of vascular malformations, including venous malformations (VM) and arteriovenous malformations (AVM). The procedure will be conducted under ultrasound guidance, and MRI will be used to assess lesion size and symptom improvement at preoperative and postoperative time points.
  Interventions: Device: Microwave Ablation

INTERVENTIONS:
Device: Microwave Ablation — This intervention involves the use of a microwave ablation catheter to treat vascular malformations, including venous malformations (VM) and arteriovenous malformations (AVM). The procedure is minimally invasive and performed under local anesthesia, with the lesion targeted using ultrasound guidance. Post-procedure imaging with MRI will be used to assess lesion size reduction and symptom improvement at several time points (preoperative, 1 month, 3 months, 6 months, and 12 months).

SUMMARY:
This clinical trial aims to assess the safety and efficacy of microwave ablation in treating vascular malformations, including both venous malformations (VM) and arteriovenous malformations (AVM). Vascular malformations are abnormal clusters of blood vessels that can cause pain, swelling, and functional impairment, significantly affecting a patient's quality of life. Microwave ablation is a minimally invasive treatment that uses heat to shrink abnormal vessels, but its effectiveness and safety for these conditions need further investigation.

The trial will enroll 150 patients (100 with venous malformations and 50 with arteriovenous malformations), all of whom will undergo a single session of microwave ablation. Ultrasound guidance will be used during the procedure to precisely target the lesions, while MRI will be used for both preoperative and postoperative evaluations to assess lesion size and track changes over time.

The primary goals of the study are to determine whether microwave ablation can reduce lesion size and improve symptoms such as pain and swelling. Additionally, the study will monitor adverse events to evaluate the safety of the procedure, including any potential complications like infection, bleeding, or nerve injury.

Patients will be followed for 12 months, with MRI scans taken at 1 month, 3 months, 6 months, and 12 months after the procedure to evaluate lesion shrinkage and monitor for any recurrence. Clinical symptoms will also be assessed at these time points to track improvement.

This study could provide important data on the safety and efficacy of microwave ablation, potentially offering a less invasive treatment option for patients with vascular malformations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinically diagnosed vascular malformations (venous malformations (VM) or arteriovenous malformations (AVM)) confirmed by MRI or ultrasound.
2. Presence of symptomatic lesions (pain, swelling, functional impairment, or ulceration) that require treatment.
3. Lesions that are amenable to microwave ablation based on preoperative clinical and imaging assessment.
4. Ability to provide informed consent or parental consent for minors (if applicable).

Exclusion Criteria:

1. Capillary malformations or congenital arteriovenous fistula.
2. Lesions that are too close to critical structures (e.g., major blood vessels or nerves) and cannot be safely treated.
3. Pregnancy or breastfeeding.
4. Severe coagulopathy or significant bleeding disorders.
5. Active infection at the treatment site.
6. Patients with severe uncontrolled systemic disease that could interfere with treatment or recovery.
7. Recent treatments (e.g., surgery, sclerotherapy, embolization) for the same lesion within the last 6 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Lesion Volume Reduction | Preoperative, 3 months, 6 months, 12 months
  This outcome measures the reduction in the volume of vascular malformations, including both venous malformations (VM) and arteriovenous malformations (AVM), after microwave ablation. MRI will be used to assess lesion size before treatment and at 1 month, 3 months, 6 months, and 12 months post-procedure. The primary goal is to achieve a ≥50% reduction in lesion volume compared to the baseline preoperative size, indicating treatment success.
Swelling and Function Improvement (Venous Malformation Symptom Score - VMSS) | Preoperative, 1 month, 3 months, 6 months, 12 months
  This outcome evaluates the improvement in symptoms such as swelling and functional impairment caused by the vascular malformation. The Venous Malformation Symptom Score (VMSS) will be used, which includes a comprehensive assessment of symptoms like pain, swelling, and the ability to perform daily activities. The VMSS will be measured preoperatively and at follow-up visits at 1 month, 3 months, 6 months, and 12 months post-treatment. A ≥50% reduction in symptom score will be considered a significant improvement.

SECONDARY OUTCOMES:
Pain Reduction (Visual Analog Scale - VAS) | Preoperative, 1 month, 3 months, 6 months, 12 months
  This outcome evaluates the improvement in pain levels experienced by participants after undergoing microwave ablation for vascular malformations. The Visual Analog Scale (VAS) will be used to measure pain intensity, with scores recorded before the procedure and at 1 month, 3 months, 6 months, and 12 months post-treatment. A reduction of ≥2 points on the VAS will be considered a significant improvement in pain management.
Adverse Events (Incidence and Severity) | 1 month, 3 months, 6 months, 12 months
  This outcome monitors the safety of the microwave ablation procedure by tracking any adverse events (AEs) or serious adverse events (SAEs) that occur during or after treatment. Events such as infection, bleeding, nerve damage, and thrombosis will be recorded. Adverse events will be categorized based on severity (mild, moderate, severe) and relatedness to the procedure. The incidence of these events will be evaluated at 1 month, 3 months, 6 months, and 12 months post-procedure.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen J, Dou J, Han Z, Liang P. Microwave Ablation for Refractory Giant Maxillofacial Arteriovenous Malformation: A Case Report. Laryngoscope. 2023 Nov;133(11):2984-2987. doi: 10.1002/lary.30664. Epub 2023 Mar 24. PMID 36960915
- [Result] Fang MR, Wang L, Li TT, Deng XW, Li XY, Lu M. [Comparison of efficacy between ultrasound-guided microwave ablation and sclerosing agents for the treatment of head and neck venous malformations]. Zhonghua Yi Xue Za Zhi. 2025 Apr 22;105(16):1256-1261. doi: 10.3760/cma.j.cn112137-20241116-02571. Chinese. PMID 40262997
- [Result] Yin HH, Wen R, Lin P, Yang H, Hu M, Yang H. Ultrasound-guided microwave ablation of soft tissue venous malformations. J Vasc Surg Venous Lymphat Disord. 2023 May;11(3):605-609. doi: 10.1016/j.jvsv.2022.11.003. Epub 2022 Dec 24. PMID 36574903
- [Result] Wang L, Lu M, Zhuang M, Liang Y, Wang SS, Li JM. Microwave ablation with hydrodissection used for the treatment of vascular malformations: effectiveness and safety study. Front Oncol. 2024 Jun 4;14:1146972. doi: 10.3389/fonc.2024.1146972. eCollection 2024. PMID 38894863
- [Result] Huang S, Xu F, Li X, Zhang H, Chen J, Zhao Z, Zhang J, Peng L, Kong X. Efficacy of ultrasound-guided microwave ablation for vascular malformations in children. J Vasc Surg Venous Lymphat Disord. 2025 Jul;13(4):102240. doi: 10.1016/j.jvsv.2025.102240. Epub 2025 Mar 25. PMID 40147690